CLINICAL TRIAL: NCT00869336
Title: Phase 2 Study - A Randomized, Multi-Center, Double-Blind, Placebo-Controlled Duration Finding Study Evaluating the Efficacy and Safety of Two Week and Four Week Once Daily Treatment of Luliconazole Cream 1% in Patients With Tinea Pedis
Brief Title: Multicenter Study of the Efficacy and Safety of Luliconazole Cream in Tinea Pedis (Athlete's Foot)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tinea Pharmaceuticals (Industry)
Responsible Party: Tinea Pharmaceuticals, Inc., Tinea Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TP-0801
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2011-06

CONDITIONS: Tinea Pedis
Keywords: Tinea Pedis; Athlete's Foot
MeSH Terms: conditions — Tinea Pedis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Luliconazole Cream 1% - 2 wks (Experimental): Daily treatment with Luliconazole Cream 1% for 2 weeks
  Interventions: Drug: Luliconazole Cream 1% - 2 wks
- Luliconazole Cream 1% - 4 wks (Experimental): Daily treatment with Luliconazole Cream 1% for 4 weeks
  Interventions: Drug: Luliconazole Cream 1% - 4 wks
- Placebo Comparator - 2 wks (Placebo Comparator): Daily treatment with Vehicle Cream for 2 weeks
  Interventions: Drug: Placebo Comparator -2 wks
- Placebo Comparator - 4 wks (Placebo Comparator): Daily treatment with Vehicle Cream for 4 weeks
  Interventions: Drug: Placebo Comparator - 4 wks

INTERVENTIONS:
Drug: Luliconazole Cream 1% - 2 wks — Topical cream applied daily for 2 weeks
  Arms: Luliconazole Cream 1% - 2 wks
Drug: Placebo Comparator -2 wks — Placebo cream applied daily for 2 weeks
  Arms: Placebo Comparator - 2 wks
Drug: Luliconazole Cream 1% - 4 wks — Topical cream applied daily for 4 weeks
  Arms: Luliconazole Cream 1% - 4 wks
Drug: Placebo Comparator - 4 wks — Placebo cream applied daily for 4 weeks
  Arms: Placebo Comparator - 4 wks

SUMMARY:
To examine the safety and optimal duration of Luliconazole Cream 1% treatments for 14 days or 28 days to achieve "complete clearance" at 2 weeks post treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of either gender must be 12 years of age or older.
2. Subjects with a clinical diagnosis of interdigital tinea pedis on one or both feet characterized by clinical evidence of a tinea infection (at least moderate erythema, moderate scaling, and mild pruritus) based on signs and symptoms.
3. Subjects with a mycological diagnosis of interdigital tinea pedis confirmed by the detection of fungal hyphae on a microscopic KOH wet mount
4. Females of child-bearing potential must have a negative urine pregnancy test and must agree to use an effective form of contraception

Exclusion Criteria:

1. Subjects with moccasin (dry type) tinea pedis; with concomitant onychomycosis of the fingernails and/or toenails on the evaluated foot, with severe dermatophytoses, a concurrent tinea infection or bacterial skin infection on the evaluated foot;
2. Female subjects who are pregnant and/or nursing or planning a pregnancy during the course of the trial.
3. Subjects who are immunocompromised (due to disease, e.g., HIV or medications
4. Subjects with a history of intolerance or hypersensitivity to imidazole compounds or the inactive components of the cream;
5. Subjects with a life-threatening condition (e.g., autoimmune deficiency syndrome, cancer, unstable angina, or myocardial infarction) within the last 6 months.
6. Subjects using the following medications:

   1. topical antifungal agent within 30 days of the baseline visit
   2. systemic antifungals within 8 weeks of the baseline visit (8 months for oral terbinafine)
   3. topical corticosteroid in treatment area(s) within 30 days of the baseline visit.
   4. systemic corticosteroids within 30 days of the baseline visit;
   5. any other topical medicated topical treatments to the treatment area(s) within 7 days of baseline visit.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2009-03; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who achieve complete clearance at 2 weeks post treatment | Two weeks post treatment

SECONDARY OUTCOMES:
Proportion of subjects who achieve effective treatment at 2 and 4 weeks post treatment | 2 and 4 weeks post treatment

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Fridley, Minnesota
  - Portland, Oregon
  - Austin, Texas
  - College Station, Texas